CLINICAL TRIAL: NCT05097989
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Efficacy and Safety of ALXN2050 in Adult Participants With Proliferative Lupus Nephritis (LN) or Immunoglobulin A Nephropathy (IgAN)
Brief Title: Study of ALXN2050 in Proliferative Lupus Nephritis (LN) or Immunoglobulin A Nephropathy (IgAN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALXN2050-NEPH-201; 2021-001426-22 (EudraCT Number)
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Lupus Nephritis; Immunoglobulin A Nephropathy; IgAN; LN
Keywords: ALXN2050; Complement Factor D; Complement Alternative Pathway; LN; IgAN
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis, IGA | interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of treatment allocation will be observed at least until Week 50.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LN Cohort: ALXN2050 180 mg (Experimental): Participants diagnosed with LN with an active flare will receive ALXN2050 in addition to standard-of-care background therapy.
  Interventions: Drug: ALXN2050
- LN Cohort: ALXN2050 120 mg (Experimental): Participants diagnosed with LN with an active flare will receive ALXN2050 in addition to standard-of-care background therapy.
  Interventions: Drug: ALXN2050
- LN Cohort: Placebo (Placebo Comparator): Participants diagnosed with LN with an active flare will receive matched placebo in addition to standard-of-care background therapy.
  Interventions: Drug: Placebo
- IgAN Cohort: ALXN2050 180 mg (Experimental): Participants diagnosed with IgAN will receive ALXN2050 in addition to standard-of-care background therapy.
  Interventions: Drug: ALXN2050
- IgAN Cohort: ALXN2050 120 mg (Experimental): Participants diagnosed with IgAN will receive ALXN2050 in addition to standard-of-care background therapy.
  Interventions: Drug: ALXN2050
- IgAN Cohort: Placebo (Placebo Comparator): Participants diagnosed with IgAN will receive matched placebo in addition to standard-of-care background therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN2050 — Oral tablets
  Other Names: ACH-0145228 (formerly)
  Arms: IgAN Cohort: ALXN2050 120 mg; IgAN Cohort: ALXN2050 180 mg; LN Cohort: ALXN2050 120 mg; LN Cohort: ALXN2050 180 mg
Drug: Placebo — Oral tablets
  Arms: IgAN Cohort: Placebo; LN Cohort: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study of ALXN2050 (120 and 180 milligrams [mg]) in addition to background therapy consistent with the standard of care in adult participants (≥ 18 to ≤ 75 years of age) with either LN or IgAN. The study will consist of an up to 6-week Screening Period, a 26-week blinded Initial Evaluation Period, a 24-week blinded Extended Treatment Period, and an Open-label Extension (OLE) Period of up to 2 years.

Safety will be monitored throughout the study.

ELIGIBILITY:
Key Inclusion Criteria:

Both Cohorts

* Participants on sodium-glucose cotransporter-2 (SGLT 2) inhibitors (eg, empagliflozin) must be on a stable dose for ≥ 3 months with no planned change in dose during the Blinded Treatment Periods (through Week 50).

LN Cohort

* Clinical diagnosis of SLE by 2019 American College of Rheumatology and European League Against Rheumatism criteria.
* Diagnosis of 2018 Revised International Society of Nephrology/Renal Pathology Society classification (active focal or diffuse proliferative LN Class III or IV) confirmed by biopsy obtained ≤ 6 months prior to Screening or during Screening Period. Participants may co-exhibit Class V disease. Participants with de novo or relapsing disease may be eligible.
* Clinically active LN at Screening requiring/receiving immunosuppression induction treatment in the opinion of the Investigator.
* Proteinuria with UPCR ≥ 1 g/g based on one 24 hour urine collection during the Screening Period.

IgAN Cohort

* Established diagnosis of primary IgAN based on kidney biopsy obtained any time prior to or during the Screening Period.
* Mean proteinuria ≥ 1 g/day on 2 complete and valid 24 hour urine collections during the Screening Period.
* For participants with a kidney biopsy performed > 1 year prior to Screening that was used for eligibility: Presence of hematuria as defined by a positive result for blood on urine dipstick or ≥ 10 red blood cells (RBCs)/high power field (hpf) microscopy on urine sediment (documented by the local laboratory) during Screening Period. Presence of hematuria documented by the central laboratory may also be acceptable.
* Compliance with stable and optimal dose of RAS inhibitor treatment including maximum allowed or tolerated ACE inhibitor and/or ARB dose for ≥ 3 months prior to Screening with no expected change in dose during the Blinded Treatment Periods (through Week 50) (participants with established intolerance to RAS inhibitors may be included).
* Controlled and stable blood pressure (defined as < 140/90 millimeters of mercury [mmHg]) over the past 3 months prior to randomization.

Key Exclusion Criteria:

Both Cohorts

* eGFR ≤ 30 milliliters/minute/1.73 squared meters during Screening calculated by Chronic Kidney Disease Epidemiology Collaboration.
* For participants with eGFR < 45 mL/min/1.73 m2 at Screening, presence of any of the following in glomeruli on most recent kidney biopsy prior to or during the Screening

Period:

1. ≥ 50% interstitial fibrosis and tubular atrophy
2. ≥ 50% glomerular sclerosis
3. ≥ 50% active crescent formation

   * Concomitant significant renal disease other than LN or IgAN on the most recent biopsy prior to or during the Screening Period.
   * History of solid organ or bone marrow transplant, or planned transplant during the Blinded Extended Treatment Period (50 weeks).
   * Splenectomy or functional asplenia.
   * Known or suspected complement deficiency, unless attributable to underlying disease (that is, LN and IgAN).
   * Bone marrow insufficiency with absolute neutrophil count < 1.3 × 10^3/microliter; thrombocytopenia (platelet count < 50,000/cubic millimeter).

LN Cohort

* Participants who have initiated any of the following treatments for the current active LN flare:

  1. Cyclophosphamide ≤ 6 months prior to Screening
  2. CNIs ≤ 1 months prior to Screening
  3. A cumulative dose of intravenous (IV) methylprednisolone > 3 g
  4. Mycophenolate mofetil > 2 g/day (or equivalent) for ≥ 8 consecutive weeks prior to Screening
  5. Prednisone or prednisone equivalent ≥ 0.5 mg/kg/day for ≥ 8 consecutive weeks prior to Screening
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 110 mmHg) on 2 or more measurements during the Screening Period.
* Prior history or clinically active SLE-related cerebritis, seizures, stroke, or stroke syndrome requiring treatment or clinically active pericarditis
* Inability to take or tolerate the standard of care background therapies

IgAN Cohort

* Diagnosis of rapid progressive glomerulonephritis as measured by eGFR loss ≥ 30% over a period of 3 months prior to or during the Screening Period.
* Secondary etiologies of IgAN.
* Prednisone or prednisone equivalent > 20 mg/day for > 14 consecutive days or any other systemic immunosuppression for the treatment of IgAN ≤ 6 months prior to Screening
* Blood pressure of ≥ 140/90 mmHg during the Screening Period confirmed on 2 measures > 30 minutes apart.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (10):
  - Research Site, Huntsville, Alabama
  - Research Site, Loma Linda, California
  - Research Site, Northridge, California
  - Research Site, Gainesville, Florida
  - Research Site, Nampa, Idaho
  - Research Site, Des Moines, Iowa
  - Research Site, Kansas City, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Argentina (4):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
- Australia (4):
  - Research Site, Clayton
  - Research Site, Liverpool
  - Research Site, Nedlands
  - Research Site, Westmead
- Brazil (5):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Salvador
- China (3):
  - Research Site, Guangzhou
  - Research Site, McKinney
  - Research Site, Shanghai
- Germany (6):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Mainz A. Rhein
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, München
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (5):
  - Research Site, Bari
  - Research Site, Brescia
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Torino
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Torreón
- Serbia (2):
  - Research Site, Niš
  - Research Site, Novi Sad
- South Korea (3):
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Palma de Mallorca
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
- Research Site, Bangkok, Thailand
- Research Site, Istanbul, Turkey (Türkiye)
- United Kingdom (6):
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Doncaster
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN2050-NEPH-201&attachmentIdentifier=65f241f9-cb8f-42ee-97ae-be75462d581b&fileName=ALXN2050-NEPH-201_CSR_Synopsis_Redacted-v1.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the immunoglobulin A nephropathy (IgAN) cohort, a total of 61 participants were enrolled in the study and randomized. For the lupus nephritis (LN) cohort, a total of 39 participants were enrolled in the study and randomized. Two doses of ALXN2050 were administered, 120 milligrams (mg) or 180 mg, both twice daily (bid).
Groups:
- IgAN Cohort: ALXN2050 120 mg; IgAN Cohort: ALXN2050 180 mg: Participants diagnosed with IgAN received ALXN2050 in addition to standard-of-care background therapy throughout the entire study.
- IgAN Cohort: Placebo: Participants diagnosed with IgAN received matched placebo in addition to standard-of-care background therapy during the Initial Evaluation Period.
- IgAN Cohort: Placebo to ALXN2050 120 mg; IgAN Cohort: Placebo to ALXN2050 180 mg: Participants diagnosed with IgAN received matched placebo in addition to standard-of-care background therapy during the Initial Evaluation Period. Participants then received ALXN2050 in addition to standard-of-care background therapy during the Extended Treatment Period and the Open-label Extension Period.
- LN Cohort: ALXN2050 120 mg; LN Cohort: ALXN2050 180 mg: Participants diagnosed with LN with an active flare received ALXN2050 in addition to standard-of-care background therapy throughout the entire study.
- LN Cohort: Placebo: Participants diagnosed with LN with an active flare received matched placebo in addition to standard-of-care background therapy during the Initial Evaluation Period and the Extended Treatment Period.
- LN Cohort: Placebo to Standard-of-care Background Therapy: Participants diagnosed with LN with an active flare received matched placebo in addition to standard-of-care background therapy during the Initial Evaluation Period and the Extended Treatment Period. The participants then received standard-of-care background therapy only during the Open-label Extension Period.
Period: Initial Evaluation Period (26 Weeks)
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo | LN Cohort: Placebo to Standard-of-care Background Therapy
Started | 9 | 26 | 26 (At randomization, participants assigned to this group were also assigned to their study treatment for the Extended Treatment Period (ALXN2050 120 mg bid or ALXN2050 180 mg bid) in a 1:1 allocation ratio.) | 0 | 0 | 6 | 17 | 16 | 0
Received at Least 1 Dose of Study Drug | 9 | 26 | 26 | 0 | 0 | 6 | 17 | 16 | 0
Completed | 9 | 26 | 24 | 0 | 0 | 2 | 13 | 11 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 4 | 4 | 5 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extended Treatment Period (24 Weeks)
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo | LN Cohort: Placebo to Standard-of-care Background Therapy
Started | 9 | 26 | 0 (After receiving placebo during the Initial Evaluation Period, participants in this cohort received either ALXN2050 180 mg or ALXN2050 120 mg, per randomization.) | 12 (After receiving placebo during the Initial Evaluation Period, participants in this cohort received ALXN2050 120 mg, per randomization.) | 11 (After receiving placebo during the Initial Evaluation Period, participants in this cohort received ALXN2050 180 mg, per randomization. One participant discontinued the study prior to entering the Extended Treatment Period.) | 2 | 13 | 10 (One participant discontinued the study prior to entering the Extended Treatment Period.) | 0
Received at Least 1 Dose of Study Drug | 6 | 19 | 0 | 10 | 9 | 2 | 9 | 10 | 0
Completed | 5 | 14 | 0 | 8 | 6 | 2 | 6 | 6 | 0
Not Completed | 4 | 12 | 0 | 4 | 5 | 0 | 7 | 4 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 4 | 8 | 0 | 1 | 3 | 0 | 7 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Open-label Extension Period (2 Years)
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo | LN Cohort: Placebo to Standard-of-care Background Therapy
Started | 5 | 14 | 0 | 8 | 6 | 2 | 5 (One participant discontinued the study prior to entering the Open-label Extension Period.) | 0 (After receiving placebo in addition to standard-of-care background therapy during the Initial Evaluation Period and the Extended Treatment Period, participants in this cohort received standard-of-care background therapy only.) | 6 (After receiving placebo in addition to standard-of-care background therapy during the Initial Evaluation Period and the Extended Treatment Period, participants in this cohort received standard-of-care background therapy only.)
Received at Least 1 Dose of Study Drug | 4 | 11 | 0 | 5 | 4 | 1 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 14 | 0 | 8 | 6 | 2 | 5 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 4 | 12 | 0 | 8 | 5 | 2 | 5 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention.
Groups:
- LN Cohort: Placebo: Participants diagnosed with LN with an active flare received matched placebo in addition to standard-of-care background therapy during the Initial Evaluation Period and the Extended Treatment Period. The participants then received standard-of-care background therapy only during the Open-label Extension Period.
- Total: Total of all reporting groups
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo | Total
Number analyzed (Participants) | 9 | 26 | 26 | 6 | 17 | 16 | 100
Age, Customized [Number; unit: Participants]
  18 - 65 years | 9 | 24 | 25 | 6 | 17 | 16 | 97
  >65 years | 0 | 2 | 1 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 10 | 6 | 12 | 13 | 53
  Male | 6 | 17 | 16 | 0 | 5 | 3 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 2 | 9 | 7 | 34
  Not Hispanic or Latino | 4 | 20 | 21 | 4 | 8 | 9 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Asian | 2 | 5 | 5 | 3 | 3 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 1 | 3
  White | 7 | 20 | 20 | 3 | 9 | 6 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Both Cohorts: Percentage Change in Proteinuria From Baseline at Week 26
Description: Proteinuria, the presence of excess proteins in the urine, was assessed using 24-hour urine collections obtained at designated timepoints. A negative change from baseline indicated an improvement in symptoms.
Time Frame: Baseline, Week 26
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies those participants evaluable for this outcome measure, and 'Number Analyzed' signifies those participants evaluable at the specified timepoints.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 9 | 25 | 23 | 2 | 11 | 11
Percentage Change | -29.3 [-51.7 to 3.5] | -26.2 [-41.2 to -7.4] | -10.3 [-29.1 to 13.4] | -84.0 [-95.4 to -44.1] | -58.0 [-75.1 to -29.2] | -55.4 [-73.3 to -25.5]
Statistical Analysis 1: Comparison: IgAN Cohort: ALXN2050 180 mg vs IgAN Cohort: Placebo; Test type: Other; p = 0.2422, ANCOVA; Percentage Difference = -17.7, 90% CI 2-sided [-37.5 to 8.3]
Statistical Analysis 2: Comparison: LN Cohort: ALXN2050 180 mg vs LN Cohort: Placebo; Test type: Other; p = 0.8701, ANCOVA; Percentage Difference = -6.0, 90% CI 2-sided [-49.3 to 74.4]

2. Secondary Outcome: Both Cohorts: Percentage Change in Proteinuria From Baseline at Week 50
Description: as for outcome 1
Time Frame: Baseline, Week 50
Population: Full Analysis Set: all participants who have been randomized and received at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies those participants evaluable for this outcome measure, and 'Number Analyzed' signifies those participants evaluable at the specified timepoints.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 5 | 12 | 8 | 6 | 1 | 5 | 6
Percentage Change | -22.0 [-58.9 to 48.0] | -30.2 [-53.6 to 4.9] | -45.9 [-67.5 to -9.9] | -14.0 [-52.2 to 54.6] | -80.7 [-95.6 to -16.5] | -68.6 [-83.5 to -40.4] | -74.4 [-85.9 to -53.5]

3. Secondary Outcome: Both Cohorts: Percentage of Participants Achieving >30% and >50% Reduction in Proteinuria at Week 26 and Week 50 Compared to Baseline
Description: Proteinuria, the presence of excess proteins in the urine, was assessed using 24-hour urine collections obtained at designated timepoints. A reduction from baseline indicated an improvement in symptoms.
Time Frame: Week 26 and Week 50
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 9 | 26 | 25 | 9 | 9 | 4 | 14 | 11
Percentage of Participants
  Week 26: >30% Reduction: number analyzed (Participants) | 9 | 26 | 25 | 0 | 0 | 4 | 14 | 11
  Week 26: >30% Reduction | 55.6 [21.2 to 86.3] | 34.6 [17.2 to 55.7] | 16.0 [4.5 to 36.1] |  |  | 50.0 [6.8 to 93.2] | 42.9 [17.7 to 71.1] | 54.5 [23.4 to 83.3]
  Week 26: >50% Reduction: number analyzed (Participants) | 9 | 26 | 25 | 0 | 0 | 4 | 14 | 11
  Week 26: >50% Reduction | 11.1 [0.3 to 48.2] | 15.4 [4.4 to 34.9] | 8.0 [1.0 to 26.0] |  |  | 50.0 [6.8 to 93.2] | 35.7 [12.8 to 64.9] | 45.5 [16.7 to 76.6]
  Week 50: >30% Reduction: number analyzed (Participants) | 5 | 14 | 0 | 9 | 9 | 4 | 8 | 7
  Week 50: >30% Reduction | 40.0 [5.3 to 85.3] | 50.0 [23.0 to 77.0] |  | 77.8 [40.0 to 97.2] | 22.2 [2.8 to 60.0] | 25.0 [0.6 to 80.6] | 50.0 [15.7 to 84.3] | 71.4 [29.0 to 96.3]
  Week 50: >50% Reduction: number analyzed (Participants) | 5 | 14 | 0 | 9 | 9 | 4 | 8 | 7
  Week 50: >50% Reduction | 0.0 [0.0 to 52.2] | 28.6 [8.4 to 58.1] |  | 55.6 [21.2 to 86.3] | 0.0 [0.0 to 33.6] | 25.0 [0.6 to 80.6] | 50.0 [15.7 to 84.3] | 57.1 [18.4 to 90.1]

4. Secondary Outcome: Both Cohorts: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 26 and Week 50
Description: Changes in kidney function were monitored using measurements of eGFR and calculated based on the Chronic Kidney Disease Epidemiology Collaboration formula. Results are reported in milliliters/minute/1.73 meters squared (mL/min/1.73 m^2). Estimates of change from baseline are least-square means based on a mixed-effect model for repeated measures model that included change from baseline as the response variable, treatment as independent variable and adjusts for covariates of baseline and the stratification factor at randomization. An increase in eGFR in response to treatment indicated an improvement in symptoms.
Time Frame: Baseline, Week 26 and Week 50
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 9 | 25 | 12 | 11 | 2 | 11 | 11
mL/min/1.73 m^2
  Week 26 | -2.29 (2.625) | -0.47 (1.564) | -1.62 (2.248) | -0.73 (2.323) | 11.92 (12.770) | -3.76 (5.590) | 8.84 (5.780)
  Week 50: number analyzed (Participants) | 5 | 16 | 8 | 6 | 2 | 6 | 6
  Week 50 | -5.97 (4.458) | -6.03 (2.520) | -3.36 (3.587) | -0.80 (4.007) | 2.58 (13.940) | -5.65 (7.450) | 5.07 (7.280)

5. Secondary Outcome: LN Cohort: Percentage of Participants Meeting the Criteria for Complete Renal Response at Week 26 and Week 50
Description: Complete renal response was defined as a decrease in urine protein to creatinine ratio (UPCR) to ≤0.5 gram/gram (g/g), an eGFR rate >60 mL/min/1.73 m^2 or no eGFR reduction ≥20% from baseline, and no treatment failure. Treatment failure was defined as the receipt of additional standard of care therapy at any time during the study for protocol-defined renal flare, severe extrarenal systemic lupus erythematosus (SLE) flare, or suboptimal response.
Time Frame: Week 26 and Week 50
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 4 | 14 | 11
Percentage of Participants
  Week 26 | 25.0 [0.6 to 80.6] | 14.3 [1.8 to 42.8] | 9.1 [0.2 to 41.3]
  Week 50: number analyzed (Participants) | 4 | 9 | 7
  Week 50 | 0.0 [0.0 to 60.2] | 22.2 [2.8 to 60.0] | 42.9 [9.9 to 81.6]

6. Secondary Outcome: LN Cohort: Percentage of Participants Meeting the Criteria for Partial Renal Response at Week 26 and Week 50
Description: Partial renal response was defined as a decrease in UPCR ≥50% compared to baseline, an eGFR rate >60 mL/min/1.73 m^2 or no eGFR reduction ≥20% from baseline, and no treatment failure. Treatment failure was defined as the receipt of additional standard of care therapy at any time during the study for protocol-defined renal flare, severe extrarenal SLE flare, or suboptimal response.
Time Frame: Week 26 and Week 50
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 4 | 14 | 11
Percentage of Participants
  Week 26 | 25.0 [0.6 to 80.6] | 14.3 [1.8 to 42.8] | 45.5 [16.7 to 76.6]
  Week 50: number analyzed (Participants) | 4 | 9 | 7
  Week 50 | 0.01 [0.0 to 60.2] | 0.01 [0.0 to 33.6] | 28.6 [3.7 to 71.0]

7. Secondary Outcome: LN Cohort: Time to the First Occurrence of UPCR ≤0.5 g/g as Measured by a Spot Urine Sample
Description: UPCR was assessed using 24-hour urine collections obtained at designated time points. The time to the first occurrence of UPCR ≤0.5 g/g was summarized by spot urine sample analysis.
Time Frame: Up to Week 50
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 6 | 17 | 16
Weeks | 2.4 [2.1 to NA] — Values were non-estimable (insufficient number of participants with events). | NA [NA to NA] — Values were non-estimable (insufficient number of participants with events). | 12.1 [4.6 to NA] — Values were non-estimable (insufficient number of participants with events).

8. Secondary Outcome: LN Cohort: Percentage of Participants Achieving Corticosteroid Taper to 7.5 mg/Day at Weeks 12, 26, and 50
Description: A corticosteroid taper was carried out per protocol at the clinical discretion of the investigator.
Time Frame: Week 12, Week 26, And Week 50
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 3 | 15 | 14
Percentage of Participants
  Week 12 | 100 [29.2 to 100] | 100 [78.2 to 100] | 78.6 [49.2 to 95.3]
  Week 26: number analyzed (Participants) | 2 | 13 | 11
  Week 26 | 100 [15.8 to 100] | 84.6 [54.6 to 98.1] | 90.9 [58.7 to 99.8]
  Week 50: number analyzed (Participants) | 2 | 6 | 6
  Week 50 | 100 [15.8 to 100] | 83.3 [35.9 to 99.6] | 100 [54.1 to 100]

9. Secondary Outcome: LN Cohort: Percentage of Participants Experiencing a Renal Flare Through Week 50
Description: Renal flare was determined in the opinion of the investigator and additional protocol-specified criteria. For participants who achieved a complete renal response, a renal flare was the reproducible recurrence of proteinuria ≥1g/g. For all other participants, a renal flare was either of the following: a reproducible increase of serum creatinine >25% higher than baseline or above the upper limit of normal (plus additional protocol-specified criteria) or a reproducible doubling of the UPCR from a 24-hour urine collection compared with the lowest previous value obtained after the first dose of study intervention.
Time Frame: Baseline Through Week 50
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 6 | 17 | 16
Percentage of Participants | 0.0 [0.0 to 45.9] | 5.9 [0.1 to 28.7] | 6.3 [0.2 to 30.2]

10. Secondary Outcome: LN Cohort: Percentage of Participants Experiencing an Extrarenal SLE Flare Through Week 50
Description: Extrarenal SLE flare was defined as an increase in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Safety of Estrogens in Lupus Erythematosus National Assessment modification ≥4 points that was not accounted for by proteinuria, hematuria, urinary cellular casts, hypocomplementemia, or an increase in anti-double-stranded DNA antibody level. The SLEDAI-2K is an instrument that was used to assesses the disease activity of extrarenal SLE flare across 18 disease descriptors. Each descriptor carried a weighted value ranging from 1-8, with the reported score calculated as the sum of these descriptors and ranging from 0 to 85. Higher scores represent increased degrees of disease activity.
Time Frame: Baseline Through Week 50
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 6 | 17 | 16
Percentage of Participants | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 18.8 [4.0 to 45.6]

11. Secondary Outcome: LN Cohort: Percentage of Participants Meeting the Criteria for Treatment Failure Through Week 50
Description: Treatment failure was defined as the receipt of additional standard of care therapy at any time during the study for protocol-defined renal flare, severe extrarenal SLE flare, or suboptimal response.
Time Frame: Baseline through Week 50
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 6 | 17 | 16
Percentage of Participants | 0.0 [0.0 to 45.9] | 5.9 [0.1 to 28.7] | 12.5 [1.6 to 38.3]

12. Secondary Outcome: LN Cohort: Change From Baseline in Serum Albumin at Week 26 and Week 50
Description: For the determination of serum albumin, blood samples were obtained at designated time points. Results reported as grams/liter (g/L).
Time Frame: Baseline, Week 26 and Week 50
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 2 | 13 | 11
g/L
  Week 26: number analyzed (Participants) | 1 | 13 | 11
  Week 26 | 11.0 | 1.5 (5.98) | 4.1 (5.70)
  Week 50: number analyzed (Participants) | 2 | 7 | 6
  Week 50 | 3.5 (4.95) | 0.1 (5.87) | 1.0 (2.83)

13. Secondary Outcome: LN Cohort: Percentage of Participants Meeting the Criteria for Suboptimal Response Through Week 50
Description: A suboptimal response was to be determined in the opinion of the investigator in addition to the following criterion: reproducible proteinuria ≤25% decreased compared to baseline based on UPCR on a 24-hour urine collection performed by a central laboratory.
Time Frame: Baseline Through Week 50
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo
Number analyzed (Participants) | 6 | 17 | 16
Percentage of Participants | 16.7 [0.4 to 64.1] | 35.3 [14.2 to 61.7] | 18.8 [4.0 to 45.6]

14. Secondary Outcome: IgAN Cohort: Percentage of Participants Meeting the Criteria for Partial Remission at Week 26 And Week 50
Description: Partial remission was defined as mean proteinuria <1 g/24 hours, based on two valid 24-hour urine collections obtained within 2 weeks prior to the study visit.
Time Frame: Week 26 and Week 50
Population: Full Analysis Set: all participants who were randomized and received at least 1 dose of study intervention. Here, 'Number Analyzed' signifies those participants who were evaluable for this outcome measure at the specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg
Number analyzed (Participants) | 9 | 26 | 25 | 9 | 9
Percentage of Participants
  Week 26: number analyzed (Participants) | 9 | 26 | 25 | 0 | 0
  Week 26 | 22.2 [2.8 to 60.0] | 23.1 [9.0 to 43.6] | 16.0 [4.5 to 36.1] |  |
  Week 50: number analyzed (Participants) | 5 | 14 | 0 | 9 | 9
  Week 50 | 0.0 [0.0 to 52.2] | 35.7 [12.8 to 64.9] |  | 55.6 [21.2 to 86.3] | 22.2 [2.8 to 60.0]

ADVERSE EVENTS:
Time Frame: From baseline (Day 1) to end of the study (Day 813)
Description: Reported serious adverse events and other adverse events data based upon the Safety Set: all participants who received at least 1 dose of study intervention. Reported all-cause mortality data based upon the Randomized Set: all randomized participants.
Arm/Group | IgAN Cohort: ALXN2050 120 mg | IgAN Cohort: ALXN2050 180 mg | IgAN Cohort: Placebo | IgAN Cohort: Placebo to ALXN2050 120 mg | IgAN Cohort: Placebo to ALXN2050 180 mg | LN Cohort: ALXN2050 120 mg | LN Cohort: ALXN2050 180 mg | LN Cohort: Placebo | LN Cohort: Placebo to Standard-of-care Background Therapy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/26 | 0/26 | 0/13 | 0/13 | 0/6 | 1/17 | 1/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/26 | 2/26 | 1/10 | 1/9 | 1/6 | 5/17 | 2/16 | 0/6
Other Adverse Events (participants affected / at risk) | 7/9 | 17/26 | 19/26 | 4/10 | 7/9 | 5/6 | 13/17 | 13/16 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgAN Cohort: ALXN2050 120 mg (N=9) | IgAN Cohort: ALXN2050 180 mg (N=26) | IgAN Cohort: Placebo (N=26) | IgAN Cohort: Placebo to ALXN2050 120 mg (N=10) | IgAN Cohort: Placebo to ALXN2050 180 mg (N=9) | LN Cohort: ALXN2050 120 mg (N=6) | LN Cohort: ALXN2050 180 mg (N=17) | LN Cohort: Placebo (N=16) | LN Cohort: Placebo to Standard-of-care Background Therapy (N=6)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IgAN Cohort: ALXN2050 120 mg (N=9) | IgAN Cohort: ALXN2050 180 mg (N=26) | IgAN Cohort: Placebo (N=26) | IgAN Cohort: Placebo to ALXN2050 120 mg (N=10) | IgAN Cohort: Placebo to ALXN2050 180 mg (N=9) | LN Cohort: ALXN2050 120 mg (N=6) | LN Cohort: ALXN2050 180 mg (N=17) | LN Cohort: Placebo (N=16) | LN Cohort: Placebo to Standard-of-care Background Therapy (N=6)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (3) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipids abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exertional rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 2 (2) | 0 (0)
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypoaesthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0/3 (0) | 0/9 (0) | 0/10 (0) | 0 (0) | 0 (0) | 0 (0) | 0/12 (0) | 1/13 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0/3 (0) | 0/9 (0) | 0/10 (0) | 0 (0) | 0 (0) | 0 (0) | 0/12 (0) | 1/13 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diet noncompliance (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study intervention dosing and recruitment were paused, consistent with a data monitoring committee recommendation. Given the anticipated length of the dosing interruption that would have impacted data interpretation following dosing re-initiation, the sponsor decided to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT05097989/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT05097989/SAP_001.pdf